CLINICAL TRIAL: NCT03294005
Title: Clinical Prediction Thyroid Cancer With Thyroid Ultrasonography
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chwen-Tzuei Chang, Consultant, China Medical University Hospital
Other Study IDs: CMUH-ENDO2054
Record Dates: First submitted 2017-09-22; First posted 2017-09-26 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with nodular goiter: Enrolled subjects with nodular goiter had thyroid sonography and thyroidectomy from 2002 January to 2016 December in CMUH. Total enrolled subject about 2000. These subjects were confirmed by pathology. Each subject had been transverse and longitudinal views of thyroid ultrasonography with high-resolution ultrasound (7-14 MHz) (HP Image Point-HS, Toshiba SSA250, GE ,Aloka SSD-1200 and Siemens S2000) that was performed by our partners - endocrinologist in all patients. Gray scale ultrasonography was routinely performed in every subject. Color Doppler ultrasonography for blood flow and thyroid fine needle aspiration was not absolute done in routine procedure. All data at least was interpreted by 3 endocrinologists under the blind method. Each subject was analyzed under thyroid echogenicity, margin, calcification, inclusion, grooving change and size & ratio size of tall and transverse.
  Interventions: Diagnostic Test: Thyroid ultrasonography

INTERVENTIONS:
Diagnostic Test: Thyroid ultrasonography — Each subject had been transverse and longitudinal views of thyroid ultrasonography with high-resolution ultrasound (7-14 MHz) (HP Image Point-HS, Toshiba SSA250, GE ,Aloka SSD-1200 and Siemens S2000) that was performed by our partners - endocrinologist in all patients.

SUMMARY:
Iodine ingestion insufficiency was widespread existence in the 50's in Taiwan, induced the hypothyroidism with the popular name "the big neck". After many experts study and evaluation, goiter was gradually disappeared after salt adding iodine in the 60's. But the nodule of the thyroid gland was widespread on the Taiwan island. This situation was a particular victim in living in the mountainous area inhabitant. The middle area populaces suffer from the thyroid gland disease really popular than other areas. Recently literature reported that the cancer rate of thyroid gland rises gradually. In according to the statistics, thyroid cancer prevalence probably has 10% in the nodular goiter.

The major early preliminary diagnosis of the thyroid cancer is thyroid fine-needle aspiration cytology (FNAC), but this technique must to have skilled clinical puncture's doctor and to have special training cytological pathology doctor. Therefore, if we can have simple fast screening tool and can make up this insufficiency, then we can achieved the fast diagnosis, rapid processing, the promotion diagnosis and treatment quality and promotes the survival percentage. The thyroid ultrasonography (Thyroid US) is one universal, fast, cheap, and the simple diagnosis nodular goiter tool. If we can friendly use this tool, we can early diagnosis & management this disease.

This research collect subjects from Jan 2002 to Dec 2016 under procedure of thyroid US, FNAC and thyroidectomy. Preliminary design index of thyroid gland tumor score (TTS) was to survey and analysis.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with nodular goiter had thyroidectomy from 2002 January to 2016 December in CMUH.
* 2. Patients had thyroid sonography within one year before thyroidectomy.
* 3. All data at least was interpreted by 3 endocrinologists under the blind method.

Exclusion Criteria:

* 1. Patients with nodular goiter hadn't thyroidectomy.
* 2. Patients hadn't thyroid sonography.
* 3. All data was interpreted by endocrinologists under the blind method, but interpretation results were inconsistent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolled subjects with nodular goiter had thyroid sonography and thyroidectomy from 2002 January to 2016 December in CMUH.
Sampling Method: Probability Sample
Enrollment: 1949 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Accuracy with (TP+TN)/(TP+TN+FP+TN) | Jun 2018

SECONDARY OUTCOMES:
Sensitivity with TP/(TP+FN) | Jun 2018
Specificity with TN/(TN+FP) | Jun 2018
Positive predictive value (PPV) with TP/(TP+FP) | Jun 2018
Negative predictive value (NPV) with TN/(TN+FN) | Jun 2018

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No